CLINICAL TRIAL: NCT04764084
Title: A Single Arm, Single Center, Phase I Trial of Niraparib Plus Anlotinib in Advanced Solid Tumors With Homologous Recombination Repair (HRR) Gene Mutations
Brief Title: Niraparib Combined With Anlotinib in Homologous Recombination Repair (HRR) Gene-mutated Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Li Huiping, Department of Breast Oncology, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-2306-912 ALTER-OC-02
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: HER2-negative Breast Cancer; Gastric Adenocarcinoma; Cholangiocarcinoma; Pancreatic Cancer
Keywords: Niraprib; Anlotinib; Homologous Recombination Repair; breast cancer; gastric Adenocarcinoma; cholangiocarcinoma; pancreatic cancer
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms; Breast Neoplasms | interventions — niraparib; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Niraparib-Anlotinib combination therapy
  Interventions: Drug: Niraparib; Drug: Anlotinib

INTERVENTIONS:
Drug: Niraparib — Niraparib 100mg or 200mg, PO, qd，d1-d21
  Other Names: Zejula
Drug: Anlotinib — Anlotinib 12mg, PO, qd，d1-d14

SUMMARY:
Homologous Recombination Repair (HRR) gene mutations can be detected in many solid tumors, patients with HRR gene mutations may benefit from PARP inhibitor. Antiangiogenic drugs can induce hypoxia and increase the sensitivity to PARP inhibitor. The combination of PARP inhibitor and antiangiogenic drug can play a synergistic anti-tumor role and achieve good efficacy in HRR gene-mutated tumors. The purpose of the study is to determine the dose limiting toxicity (DLT) and maximum tolerable dose (MTD) of Niraparib plus Anlotinib in HRR gene-mutated advanced solid tumors, and evaluate the safety and effectiveness of this combination therapy preliminarily.

DETAILED DESCRIPTION:
This is a single-arm, single-center, phase I study to investigate the DLT and MDT, safety and efficacy of Niraparib combined with Anlotinib in the treatment of advanced solid tumors with HRR gene mutations. In this study, 52 histological or cytological diagnosis, previous treatment failure patients of HER2 negative breast cancer, cholangiocarcinoma, gastric adenocarcinoma and pancreatic cancer are included and receive Niraparib combined with Anlotinib. Patients are required to carry pathogenic or suspected pathogenic gBRCA or sBRCA mutations, or HRR gene mutations defined by the inclusion criteria. The study will be divided into two phase. The first phase will include 6-12 patients on a 21-day cycle to determine the DLT and MTD. In the second phase, 40 patients will be included to treated with Niraparib plus Anlotinib until disease progression or intolerable toxicity or withdrawal of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects understand the trial process, sign informed consent, agree to participate in the study, and have the ability to follow the protocol;
* 18 ~ 70 years old
* HER2 negative breast cancer, cholangiocarcinoma, gastric adenocarcinoma and pancreatic cancer confirmed by histology or cytology meet any of the following conditions: first line treatment failure of HER2 negative breast cancer; first line treatment failure of cholangiocarcinoma; second line treatment failure of gastric adenocarcinoma; first line treatment failure of pancreatic cancer
* At least one measurable target lesion that meet RECIST 1.1 criteria
* Can provide paraffin-embedded tumor tissue samples or plasma samples for HRR gene detection
* Carry pathogenic or suspected pathogenic germline or somatic HRR gene mutations, HRR genes include BRCA1, BRCA2, ATM, ATR, BAP1, BRIP1, CHEK2, FANCA, PALB2 and RAD51, mutations in other HRR genes should be evaluated by researchers and the pathogenicity should be supported by published literature or clinical studies.
* ECOG physical status score is 0-1
* Life expectancy > 6 months
* Good organ function, including: Neutrophil count >= 1500 / μL; Platelets >= 100,000 / μL; Hemoglobin >= 10g / dL; Serum creatinine <= 1.5 times the upper limit of normal value, or creatinine clearance >= 60mL / min (calculated according to Cockcroft-Gault formula); Total bilirubin <= 1.5 times the upper limit of normal value or direct bilirubin <= 1.0 times the upper limit of normal value; AST and ALT <= 2.5 times the upper limit of normal value. When liver metastases are present, it must be <= 5 times the upper limit of normal value
* The toxic side effects of any previous chemotherapy have recovered to <= CTCAE level 1 or baseline levels, except for sensory neuropathy or hair loss with stable symptoms <= CTCAE level 2

Exclusion Criteria:

* People who are known to be allergic to Niraparib or Anlotinib (or active or inactive ingredients of drugs with similar chemical structure)
* Symptomatic, uncontrolled brain or pia mater metastases
* Underwent major surgery within 3 weeks before the study began or has not recovered after surgery
* Received palliative radiotherapy of > 20% bone marrow 1 week before enrollment
* Have invasive cancer other than ovarian cancer (except fully treated basal or squamous cell skin cancer) within 2 years before enrollment
* Patients with tumor invasion of large vessels
* Previous or currently diagnosed myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Severe or uncontrolled diseases, including but not limited to: uncontrollable nausea and vomiting, inability to swallow or gastrointestinal diseases that may interfere with drug absorption and metabolism; active viral infections; mental illnesses that affect patients' signed informed consent History of bleeding tendency and thrombosis; history of severe cardiovascular disease
* Laboratory abnormalities: hyponatremia; hypokalemia; uncontrollable nail function abnormalities
* Receive platelet or red blood cell transfusions within 4 weeks
* Patients who are pregnant or nursing, or who plan to become pregnant during study treatment
* Have previously received any PARP inhibitor or Anlotinib treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) and maximum tolerated dose (MTD) | 4 weeks

SECONDARY OUTCOMES:
The frequency and severity of adverse events | Baseline through 1 year
  The frequency and severity of adverse events and toxicity based upon NCI CTCAE version 5.0 during subjects receiving the treatment
Objective Response Rate (ORR) | at 6 months
  The ORR is a combination of CR (the target lesion completely disappeared over 4 weeks) and PR (Target lesions were reduced by more than 30% for more than 4 weeks).
Progression-free survival (PFS) | at 6 months
  PFS is defined as the time from enrollment to first documentation of tumor progression, or to death due to any cause in the absence of previous documentation of objective tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Li, M.D., Principal Investigator — Peking University Cancer Hospital & Institute; Jiafu Ji, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Within six months after the trial complete, study protocol, informed consent form and clinical study report will be shared.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Within six months after the trial complete
Access Criteria: Publication